CLINICAL TRIAL: NCT05372432
Title: Hand Dominance in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Lecturer Doctor, Ufuk University
Other Study IDs: 2021-04-05
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Handgrip strengths measurements with Jamar-type hand dynamometer and, tip pinch strengths measurements with pinchmeter — The handgrip strength and tip pinch strength of the participants were measured using the Jamar-type hand dynamometer and pinch meter available in our clinic. The handgrip strengths were measured with shoulders in adduction and neutral rotation, elbows in 90 degrees flexion, and forearms and wrists in a neutral position, while the tip pinch strengths were measured by squeezing a pinch meter between the thumb and index finger. Participants took a deep breath and then applied gripping force with maximal force while exhaling. In the analysis, the average of the three measurements made with an interval of five minutes was taken as the basis for the analysis.
Other: The Nine Hole Peg Test — This test was used to evaluate the hand dexterity of the participants. This test consists of a square area and nine holes in this area, nine cylinders suitable for these holes, and a storage box. Participants quickly took the nine cylinders from the storage box and placed them in the holes, and after placing all the cylinders, they put the cylinders back in the storage box one by one. In the evaluation of the test, the time elapsed during these operations was measured in seconds with a chronometer, and shorter times were considered to indicate better hand dexterity.

SUMMARY:
Evaluating laterality changes in different psychiatric and neurodevelopmental diseases has recently been one of the popular perspectives of laterality studies. There are studies reporting changes in functional and structural hemispheric asymmetries in some neurodevelopmental and psychiatric diseases, and thus relations with atypical lateralization patterns or handedness. There is no study in the literature evaluating brain lateralization or handedness in fibromyalgia. The aim of our study is to evaluate the relationship between handedness, which is an indicator of brain lateralization, and fibromyalgia disease severity and functional outcomes related to fibromyalgia in patients with fibromyalgia. This cross-sectional study included 40 fibromyalgia patients aged 20-50 years, meeting the American College of Rheumatology 2016 Fibromyalgia Diagnostic Criteria, and 40 healthy volunteers in the same age range as the control group. Information about the age, gender, height, weight, and comorbidities of the participants included in the study were recorded. In addition, information about the duration of fibromyalgia diagnosis and pharmacological and non-pharmacological treatments for fibromyalgia were also recorded in the patient group.

Handgrip strengths with Jamar-type hand dynamometer, tip pinch strengths with pinch meter, and hand dexterities with the Nine-Hole Peg Test were evaluated for both hands of all participants. The Edinburgh Handedness Inventory, Beck Depression Inventory, and Beck Anxiety Inventory were administered to all participants. In addition, the American College of Rheumatology 2016 Fibromyalgia Diagnostic Criteria was questioned in the patient group, and the Revised Fibromyalgia Impact Questionnaire was applied.

ELIGIBILITY:
Inclusion Criteria:

* This study included 40 fibromyalgia patients aged 20-50 years, meeting the American College of Rheumatology (ACR) 2016 Fibromyalgia Diagnostic Criteria.

Exclusion Criteria:

* Exclusion criteria were defined as being younger than 20 years of age, older than 50 years of age, having systemic, inflammatory, degenerative, and neurological diseases that may lead to loss of hand and finger grip strength and dexterity, and a history of hand surgery or trauma in the last three months.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This cross-sectional study included 40 fibromyalgia patients aged 20-50 years, meeting the American College of Rheumatology (ACR) 2016 Fibromyalgia Diagnostic Criteria, and 40 healthy volunteers in the same age range as the control group.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
The handgrip and tip pinch strengths | 6 months
  The handgrip strength and tip pinch strength of the participants were measured using the Jamar-type hand dynamometer and pinch meter available in our clinic. In the analysis, the average of the three measurements made with an interval of five minutes was taken as the basis for the analysis.
The Nine Hole Peg Test | 6 months
  This test was used to evaluate the hand dexterity of the participants. This test consists of a square area and nine holes in this area, nine cylinders suitable for these holes, and a storage box. Participants quickly took the nine cylinders from the storage box and placed them in the holes, and after placing all the cylinders, they put the cylinders back in the storage box one by one. The shorter test times were considered to indicate better hand dexterity.
The Edinburgh Handedness Inventory | 6 months
  It is a questionnaire developed by Oldfield in 1971 to evaluate handedness. This inventory questions individuals' hand use in 10 different activities of daily living (writing, drawing, throwing, using scissors, brushing teeth, using a knife, using a spoon, using a broom, lighting a match, opening a box). In the inventory, there are two boxes for each activity questioning the use of the right and left hand. Only the right or left hand is always used for the specified activity; if the other hand is not used at all, both boxes for the used hand are checked. Generally, if the right or left hand is used for the specified activity, one of the boxes for the used hand is checked. If the specified activity is performed using both hands, one of the boxes on both the right and the left is checked. Right, and left-hand scores are calculated by counting the boxes checked for right and left-hand use.

SECONDARY OUTCOMES:
Beck Depression Inventory | 6 months
  This scale evaluates the level and severity of depressive symptoms. The scale consists of 21 questions in a 4-point Likert structure, where each question is scored between 0 and 3. Higher scores indicate higher levels of depression.
Beck Anxiety Inventory | 6 months
  This scale determines the frequency of anxiety symptoms experienced by individuals. The scale consists of 21 questions in a 4-point Likert structure, where each question is scored between 0 and 3. Higher scores indicate more severe anxiety.
The American College of Rheumatology 2016 Fibromyalgia Diagnostic Criteria | 6 months
  It is a set of diagnostic criteria developed for the diagnosis of fibromyalgia and created as a result of the revision of previously used diagnostic criteria. It consists of two parts, the widespread pain index (WPI) and the symptom severity scale (SSS). In the evaluation of the Fibromyalgia Severity Scale (FSS), WPI and SSS scores are collected. The total score ranges from 12 to 31. A higher score indicates greater disease severity. WPI ≥7 and SSS score ≥5, or WPI=4-6 and SSS score ≥9 suggest a diagnosis of fibromyalgia.
The Revised Fibromyalgia Impact Questionnaire | 6 months
  This questionnaire evaluates functional limitations and disability due to fibromyalgia. The questionnaire, which consists of 21 questions in total, consists of three parts: function, overall impact, and symptoms. The answers to each question are marked on a scale from 0 to 10. The total score is calculated by summing the results by dividing the score of the first section by three, the score of the second section by one, and the score of the third section by two. Higher scores indicate a more fibromyalgia-related disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No